CLINICAL TRIAL: NCT06517810
Title: Pediatric Selective Cytopheretic Device (SCD-PED, QUELIMMUNE) for Critically Ill Children With Acute Kidney Injury: A Humanitarian Device Exemption (HDE) Surveillance Registry Protocol
Brief Title: QUELIMMUNE (SCD-PED) PediAtric SurVeillance REgistry
Acronym: SAVE
Status: Recruiting | Type: Observational
Sponsor: SeaStar Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: SCD-PED-HDE-1
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-04

CONDITIONS: Acute Kidney Injury; Acute Kidney Injury Due to Sepsis
Keywords: continuous kidney replacement therapy; continuous renal replacement therapy; acute kidney injury; organ failure; inflammation; dialysis
MeSH Terms: conditions — Acute Kidney Injury; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- QUELIMMUNE Surveillance Registry Participants: All patients treated with the QUELIMMUNE device as a part of clinical practice under the approved HDE indication must be included in this registry.
  Interventions: Device: QUELIMMUNE (SCD-PED)

INTERVENTIONS:
Device: QUELIMMUNE (SCD-PED) — QUELIMMUNE device used as part of clinical practice.

SUMMARY:
QUELIMMUNE is FDA-approved under an HDE for the treatment of pediatric patients (weight ≥10kg and age ≤22 years) with AKI due to sepsis or a septic condition on antibiotic therapy and requiring RRT.

The purpose of this surveillance registry is to prospectively collect safety data among all patients treated with QUELIMMUNE under the HDE. More specifically, we intend on comparing the incidence of new (secondary) blood stream infections in the first 28 days after SCD-PED initiation to a comparator group of matched CKRT patients with sepsis who did not receive treatment with QUELIMMUNE

ELIGIBILITY:
Inclusion Criteria:

* All patients initiated on QUELIMMUNE therapy under the HDE-approved indication

Exclusion Criteria:

* Weight <10kg
* Age >22 years
* Known allergy to any components of QUELIMMUNE

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients (weight ≥10kg and age ≤22 years) with acute kidney injury (AKI) due to sepsis or a septic condition on antibiotic therapy and requiring renal replacement therapy (RRT), per device Instructions For Use. All patients who receive treatment with QUELIMMUNE as part of their therapy are included in this registry.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Safety | 28 days or through hospital discharge, whichever is sooner
  New (secondary) bloodstream infections within 28 days from the time of QUELIMMUNE initiation or through hospital discharge, whichever is sooner

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Children's of Alabama, Birmingham, Alabama
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - UCSF Benioff Children's, San Francisco, California
  - Children's Hospital of Atlanta - Arthur M. Blank, Atlanta, Georgia
  - Children's Hospital of Atlanta - Scottish Rite, Atlanta, Georgia
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - CS Mott Children's Hospital, Ann Arbor, Michigan
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Cleveland Clinic Children's Hospital, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Medical Center Dallas, Dallas, Texas
  - Cook Children's Hospital, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No